CLINICAL TRIAL: NCT06729788
Title: Evaluation of Resin Infiltrate As Pit and Fissure Sealant in Permanent Molars (In Vivo& in Vitro)
Brief Title: Resin Infiltrate As Pit and Fissure Sealant in Permanent Molars
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Salsabeel Mahmoud Abdelgaffar Shalaby, Dentist, Pediatric dentistry, Oral Health and Preventive Dentistry Department, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Resin Infiltrate
Record Dates: First submitted 2024-12-04; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Resin Infiltration; Pit and Fissure Sealant; Permanent Molars
MeSH Terms: conditions — Van der Woude syndrome | interventions — In Vitro Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For the application of ICON, The cleaned fissure was etched using an Icon-Etch in its special syringe for 2 minutes. Then the tooth was rinsed off using water for at least 30 seconds and dried with oil-free and water-free air. Followed by application of the Icon-Dry applied into the fissure and let sit for 30 seconds. The excess of the Icon-Dry was removed and dried with oil-free and water-free air.an ample amount of Icon-Infiltrate is applied into the fissure away from the direct light of the dental unit and let sit for 3 minutes. After excess removal, it will be cured with a light source* according to the manufacturer's instructions. A second layer of the Icon Infiltrate was applied and cured in the same way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- ICON resin infiltration group (in vivo) (Experimental): The fissure of selected teeth will be sealed with ICON resin infiltration Material (DMG Dental UK)
  Interventions: Drug: ICON resin infiltration Material group in vivo
- Resin-based fissure sealant group (in vivo) (Placebo Comparator): The fissure of selected teeth will be sealed with resin-based fissure sealant (Heliosael)
  Interventions: Drug: Resin-based fissure sealant group in vivo
- ICON resin infiltration Material (in vitro) (Experimental): The fissure of selected teeth will be sealed with ICON resin infiltration Material (DMG Dental UK)
  Interventions: Drug: ICON resin infiltration in vitro
- Resin-based fissure sealant (in vitro) (Placebo Comparator): The fissure of selected teeth will be sealed with resin-based fissure sealant (Heliosael)**
  Interventions: Drug: Resin-based fissure sealant in vitro

INTERVENTIONS:
Drug: ICON resin infiltration Material group in vivo — The fissure of selected teeth will be sealed with ICON resin infiltration Material (DMG Dental UK).
  Arms: ICON resin infiltration group (in vivo)
Drug: Resin-based fissure sealant group in vivo — The fissure of selected teeth will be sealed with resin-based fissure sealant (Heliosael)
  Arms: Resin-based fissure sealant group (in vivo)
Drug: ICON resin infiltration in vitro — The fissure of selected teeth will be sealed with ICON resin infiltration Material (DMG Dental UK) in vitro
  Arms: ICON resin infiltration Material (in vitro)
Drug: Resin-based fissure sealant in vitro — The fissure of selected teeth will be sealed with resin-based fissure sealant (Heliosael) in vitro
  Arms: Resin-based fissure sealant (in vitro)

SUMMARY:
The aim of this study is to evaluate and compare the clinical effectiveness of ICON resin Infiltration versus conventional sealant and the microleakage and penetration depth of the two sealant materials.

DETAILED DESCRIPTION:
Using the resin infiltration technique as a different approach for sealing pits and fissures creates a diffusion barrier as resin infiltrate tends to inhibit enamel pores that serve as diffusion channels for acids and dissolved minerals within the lesion body. A low-viscosity resin that can penetrate into caries lesions, which is referred to as resin infiltration technique. The mechanisms associated with this method depend on the infiltration of subsurface lesions with low-viscosity light-curing resins after eroding the highly mineralized surface layer and increasing penetration depth. This method is believed to overcome the limitations of sealant applications and is considered to be a better alternative for the treatment of initial caries lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the children from 6 to 8 years.
2. Healthy children free from any systemic disease.
3. Show bilaterally sound fully erupted lower first permanent molars with deep narrow central fissures and supplemental grooves.
4. The eruption time of these molars should not exceed 3 years.
5. No sign of pain or active periodontal disease in the selected teeth.

Exclusion Criteria:

1. Children with fillings or sealants in the selected teeth.
2. Children with clinical evidence of caries in the selected teeth either white spot lesions or cavities.
3. Children with an allergy to any drug, such as resin restorative material.
4. Children with Extremely poor oral hygiene.
5. Hypoplastic teeth.
6. Children with bruxism.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2025-01-04 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical effectiveness of ICON resin and the sealant retention using Simonsen's criteria. | 3 minutes for application of ICON. The children will be recalled at 3, 6, and 9 months
  172 permanent mandibular molars out of 86 children will be randomly allocated into two equal groups. Group 1: The fissure of selected teeth will be sealed with ICON resin infiltration Material (DMG Dental UK). Group 2: The fissure of selected teeth will be sealed with resin-based fissure sealant (Heliosael).For application of ICON, an ample amount of Icon-Infiltrate is applied into the fissure away from the direct light of the dental unit and let sit for 3 minutes. After excess removal, it will be cured with a light source. A second layer of the Icon Infiltrate was applied and cured in the same way. For Heliosael application, The sealant will be carefully applied starting from the maximum depth of the central ﬁssure up towards two. Sealant retention will be evaluated using Simonsen's criteria. (Completely present: no sealant ledge is present, Partially present: part of the sealed pit or fissure, Complete missing: no sealant ledge is present.

SECONDARY OUTCOMES:
Evaluate and compare the microleakage and penetration depth of the two sealant materials | thirty seconds for application of Heliosael.The children will be recalled at 3, 6, and 9 months
  20 teeth will be randomly assigned into two equal experimental groups . Experimental Group I: The fissure of selected teeth will be sealed with ICON resin infiltration. Experimental Group II: The fissure of selected teeth will be sealed with resin-based fissure sealant (Heliosael).
  After removal from the dye teeth will be rinsed with water, cleaned, and sectioned longitudinally through the center of the restorations in a buccolingual direction with a double-sided diamond disc and will be given a code number to permit blind evaluation. For each specimen, the dye penetration along the buccal and lingual margins on each sectioned surface will be digitally photographed at 10x under a stereomicroscope. The degree of microleakage was scored by a single observer.

CONTACTS AND LOCATIONS:
Locations (1):
- Salsabeel M Abdelgaffar, Tanta, ELGharbia, Egypt

REFERENCES:
- [Background] Lam PPY, Sardana D, Ekambaram M, Lee GHM, Yiu CKY. Effectiveness of Pit and Fissure Sealants for Preventing and Arresting Occlusal Caries in Primary Molars: A Systematic Review and Meta-Analysis. J Evid Based Dent Pract. 2020 Jun;20(2):101404. doi: 10.1016/j.jebdp.2020.101404. Epub 2020 Jan 29. PMID 32473795